CLINICAL TRIAL: NCT02172352
Title: Dose Ranging Study of Ba 679 BR Inhalation Powder Following Single Inhalation in COPD Patients - Double-blind, Placebo-controlled, 4 Treatment, 4 Period Crossover Study-
Brief Title: Dose Ranging Study of Ba 679 BR Inhalation Powder in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.139
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

ARMS (4):
- Ba 679 BR low dose (Experimental)
  Interventions: Drug: Ba 679 BR low dose
- Placebo inhalation powder (Placebo Comparator)
  Interventions: Drug: Placebo inhalation powder
- Ba 679 BR middle dose (Experimental)
  Interventions: Drug: Ba 679 BR middle dose
- Ba 679 BR high dose (Experimental)
  Interventions: Drug: Ba 679 BR high dose

INTERVENTIONS:
Drug: Ba 679 BR low dose
  Arms: Ba 679 BR low dose
Drug: Ba 679 BR middle dose
  Arms: Ba 679 BR middle dose
Drug: Ba 679 BR high dose
  Arms: Ba 679 BR high dose
Drug: Placebo inhalation powder
  Arms: Placebo inhalation powder

SUMMARY:
To investigate the dose response following single inhalation of Ba 679 BR inhalation powder in COPD patients using pulmonary functions as indicators, and to compare data obtained with overseas study findings

ELIGIBILITY:
Inclusion Criteria:

1. In a pulmonary function test of Screening Test II, FEV1.0 was less than 70% of predict normal and FEV1.0 was less than 70% of FVC.
2. In the reversibility test of Screening Test II, FEV1.0 was improved by 10% or more at 1 hour after inhalation of 2 puffs of an anticholinergic agent (Tersigan ® Aerozol)
3. History of smoking (< no. of cigarettes a day x no. of years of smoking > = 200 or more)
4. 40 years of age or older
5. Regardless of sex and the length of disease period

Exclusion Criteria:

1. A history of bronchial asthma
2. A history of atopic disease, such as allergic rhinitis
3. Blood eosinophil of 440/µl or more
4. Continuous use of steroid drugs (oral administration, inhalation or injection) at a dose equivalent to over 5 mg daily of prednisolone
5. A history of respiratory infection, including virus infection within 1 month before study initiation
6. Tuberculosis, lung cancer or a history of pneumonectomy
7. Glaucoma
8. Under treatment of benign prostatic hypertrophy
9. Hypersensitivity to anticholinergic agents or sympathomimetics
10. Difficulty in expectoration of sputum
11. Serious heart disease, renal disease, hepatic disease, endocrine disease or metabolic disease
12. Use of any β blockers
13. A history of myocardial infarction within the past 1 year
14. A history of heart failure, cor pulmonale or arrhythmia requiring medication within the past 3 years
15. A history of drug abuse or alcoholism
16. Treatment of psychotic disease
17. Pregnancy, possible pregnancy or lactation
18. A history of participation in any other clinical studies within the past 6 months
19. Judgment by the investigator that the patient is ineligible for inclusion in the present study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 1998-07; Primary Completion 1999-05 (Actual)

PRIMARY OUTCOMES:
FEV1.0 max (maximum forced expiratory volume in one second) | before and up to 24 hours after each study drug administration

SECONDARY OUTCOMES:
FEV1.0 AUC 0-24 (forced expiratory volume in one second as area under the curve 0 to 24 hours after administration) | before and up to 24 hours after each study drug administration
FEV1.0 time to response | before and up to 24 hours after each study drug administration
FEV1.0 Tmax (time to FEV1.0 max) | before and up to 24 hours after each study drug administration
FEV1.0 at measuring time points up to 24 hours after administration of study drug | before and up to 24 hours after each study drug administration
FVC AUC 0-24 (forced vital capacity as area under the curve 0 to 24 hours after administration) | before and up to 24 hours after each study drug administration
FVC max | before and up to 24 hours after each study drug administration
FVC at measuring time points up to 24 hours after administration of study drug | before and up to 24 hours after each study drug administration
Occurrence of adverse events | up to 29 days
Changes in blood pressure | before and up to 24 hours after each study drug administration
Changes in pulse rate | before and up to 24 hours after each study drug administration
Changes in transdermal O2 saturation | before and up to 24 hours after each study drug administration
Abnormal findings in electrocardiogram (ECG) | before and 1.5 and 24 hours after each administration of study drug
Abnormal changes in laboratory measurements | at 24 hours after last study drug administration
Urinary excretion rate | before (from 4 hours pre-dosing until immediately before dosing) and 0-2, 2-4, 4-8, 8-12 and 12-24 hours after drug administration
MMEF AUC 0-24 (maximal midexpiratory flow as area under the curve 0 to 24 hours after administration) | before and up to 24 hours after each study drug administration
MMEF max | before and up to 24 hours after each study drug administration
MMEF at measuring time points up to 24 hours after administration of study drug | before and up to 24 hours after each study drug administration